CLINICAL TRIAL: NCT06076928
Title: Brain Computer Interface (BCI) Integrated Wearable Hand Robotic Glove System for Upper Limb Stroke Rehabilitation: A 3-arm Randomized Controlled Trial
Brief Title: Brain Computer Interface (BCI) Integrated Wearable Hand Robotic Glove System for Upper Limb Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other); Singapore University of Technology & Design (Unknown); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB 2022/00694
Record Dates: First submitted 2023-09-20; First posted 2023-10-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Brain Computer Interface; Hand exoskeleton robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study design is a prospective, single-centre, single blinded 3-arm randomised controlled trial to compare upper extremity motor and functional outcomes and health related quality of life (HR-QOL) of 3 treatment modalities which are fully clinic-based and supervised by trained occupational therapists (OT). Participants will undergo dose matched training interventions with 1:1 allocation using single-blinded RCT.
Who Masked: Outcomes Assessor
Masking Description: Assessors (occupational therapist performing measurements/outcome) not involved in participant training will be blinded to assignments of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional supervised occupational therapy (CT) (Sham Comparator): CT consists of standard occupational therapy for hand function which includes but not limited to the following treatment (1) passive and active mobilisation; (2) spasticity management; (3) training with use of various modalities/equipment; (4) gross and fine motor training including reach and grasp/release functions, and object manipulation; (5) grasp training: cylindrical, spherical, intrinsic, 2-finger pincer and 3-finger grip.
  Interventions: Other: Standard Treatment of Care
- HandyRehab (HR) with supervised training by OT (Active Comparator): HR training consists of (1) passive and active mobilisation (2) spasticity management (3) gross motor training with HR applied (4) grasp training: cylindrical, spherical, intrinsic, 2-finger pincer and 3-finger grip.
  Interventions: Device: HandyRehab (HR); Other: Standard Treatment of Care
- HandyRehab integrated with BCI (BCI-HR) with supervised training by OT (Experimental): BCI-HR training consists of (1) passive and active mobilisation (2) spasticity management (3) gross motor training with BCI-HR applied (4) grasp training: cylindrical, spherical, intrinsic, 2-finger pincer and 3-finger grip.
  Interventions: Device: Brain Computer Interface integrated HandyRehab platform (BCI-HR); Other: Standard Treatment of Care

INTERVENTIONS:
Device: Brain Computer Interface integrated HandyRehab platform (BCI-HR) — To test the usability, safety and efficacy of an experimental prototype of a wearable hand robotic glove integrated with brain computer interface system being developed and researched.
  Arms: HandyRehab integrated with BCI (BCI-HR) with supervised training by OT
Device: HandyRehab (HR) — A wearable hand robotic glove approved by Health Sciences Authority, class I commercial device
  Arms: HandyRehab (HR) with supervised training by OT
Other: Standard Treatment of Care — Standard Conventional Occupational Therapy

SUMMARY:
Upper extremity (UE) recovery remains a huge rehabilitation challenge with largely incomplete recovery of the upper limb post stroke. This is due to heavier priorities placed on other stroke competencies such as mobility, activities of daily living training and home integration which results in suboptimal amounts of time spent in upper limb training post stroke.

In this study the investigators plan to pilot brain computer interface (BCI) integrated wearable hand robotic glove (HandyRehab) system for upper limb stroke rehabilitation.

DETAILED DESCRIPTION:
Robot-aided therapy have shown promising results in rehabilitation recovery in stroke patients while reducing strain and effort for both the therapist and suitable patients.

HandyRehab (HR) is a portable, wearable hand robotic glove used for functional training. The integration of Brain Computer Interface (BCI) platform with HR provides an alternative way of communication or intended movement through end-effectors for stroke and potentially facilitate neuroplasticity, improving motor functions.

This study aims to validate the usability of intensive training with HandyRehab (HR) compared with conventional occupational therapy (CT). Feasibility and safety of the novel BCI-HR will be examined and objective measures of clinical efficacy will be compared across all 3 platforms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-85 years, males and females
2. First diagnosis of stroke (ischemic or haemorrhagic), confirmed by neurologist/neurosurgeon/CT/MRI imaging
3. > 16 weeks post stroke
4. Hemiplegic pattern of post-stroke weakness
5. MRC ≥ 2/5 motor power and above for shoulder abduction & elbow flexion
6. MRC 0 to 4/5 motor power and above for finger flexors &/or extensors of thumb, index, middle fingers
7. Screening Fugl-Meyer wrist hand sub score <18/24
8. Spasticity MAS <3 for thumb, index, and middle fingers
9. Able to discriminate thumb and index sensation to pain
10. Hand sizes within 170-200mm (length) &75-85mm (width), compatible with HandyRehab robotic glove
11. BCI compatible brain states using a standardised screening protocol
12. Able to understand simple commands with Mini Mental state examination scores MMSE > 21/30)
13. Able to give informed consent

    * Subjects who are unable to clear BCI screening 11. will be randomised to either CT or HR groups.

Exclusion Criteria:

Neurological

* Recurrent stroke
* Diagnosis of neurodegenerative disease; e.g. Parkinson's' disease, Dementia, ALS

Medical:

- unstable medical or neurological conditions, life expectancy <6 months, end-organ renal failure on dialysis, severe heart failure, postural hypotension, history of uncontrolled sepsis, epilepsy with seizure within 3 months of informed consent, skin conditions which could potentially be worsened by wearable robot (ulcers, open wounds, eczema, infections etc)

Postural:

* Unable to tolerate upright posture or sit unaided for < 90min with rest breaks
* Cognitive/behavioural/visual:
* Severe dysphasia/aphasia, severe visual neglect/blindness, untreated severe depression, psychiatric illness, unable to understand study requirements

Upper limb:

* Moderate to severe spasticity (Modified Ashworth scale MAS ≥2)
* Hand/arm related pain (VAS Pain ≥ 5/10),
* Presence of finger contractures, reduced functional range of motion, limiting functional wrist/finger movements, active fractures or arthritis with deformities
* Severe limb ataxia/apraxia
* Severe post stroke hemi-anaesthesia in affected UE

BCI incompatibility:

* Motor imagery EEG signals unable to be detected
* Presence of craniectomy skull defect (affecting BCI cap fit and electrode contact)
* Concomitant participation in other interventional research trials
* Resident of nursing home or overseas country which may compromise attendance at research site
* Pregnant or lactating females will not be allowed to participate

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) Score | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Functional and dexterity score in the affected arm evaluated using 19 tests of motor function across 4 subsets; minimum score = 0, maximum score = 57, with higher score indicating better function.

SECONDARY OUTCOMES:
Fugl-Meyer Motor Assessment (FMA) scale | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Change in Fugl Meyer Motor Assessment score in the affected arm, minimum: 0, maximum: 66 with higher scores indicating greater levels of mobility function
Grip Strength (kg) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Measured by Digital hand-held Dynamometer (mean of 3 readings) for both hands
Box and Block Test (BBT) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Measures unilateral gross manual dexterity.
Nine Hole Peg Test (NHPT) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Measures finger dexterity in stroke patients.
Self-efficacy outcomes by UPSET (upper limb self-efficacy test) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Questionnaire to measure self-efficacy in various tasks after stroke.
Hr-QOL scales using SS-QOL (Stroke specific Quality of Life scale) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Quality of life scale specific to stroke patients, minimum 49, maximum 245; with higher scores indicating better function.
Patient reported Outcome Measures (PROMs) using subjective scales (Likert 0-5) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Measures patient's opinion on the usability of HR and BCI-HR
Montreal Cognitive Assessment (MOCA) | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Screening assessment to determine cognitive impairment.
Rey Auditory Verbal Learning Test (RAVLT) | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Cognitive assessment to evaluate verbal learning and memory
Trail Making Test (TMT) | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Neuropsychological test assessing visual attention and task switching.
Digit Span | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Cognitive Assessment of both forward and backward variants.
Controlled Oral Word Association Test (COWAT) | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Neuropsychological measure of verbal fluency.

OTHER OUTCOMES:
Modified Ashworth Scale (MAS) | Weeks 0 (baseline), 6 (end training), 24, 52 (follow-up)
  Measures the level of spasticity at the elbow and finger flexors of proximal interphalangeal joint regions; scored from "0 to 4" with "4" indicating affected part is more spastic in flexion/extension.
Visual Analogue Scale (self-reported pain score) | Weeks 0 (baseline), 6 (end training), 12, 24, 52 (follow-up)
  Unidimensional measure of pain intensity; "0" being no pain and "10" being worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chua, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No